CLINICAL TRIAL: NCT06403696
Title: Ultrasonography-based Prediction of Post-operative Airway Complications in Pediatric Patients
Brief Title: Predicting Post-op Airway Complications in Pediatric Patients Using Ultrasonography
Status: Completed | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Mihrican SAYAN, Specialist Doctor, Çanakkale Onsekiz Mart University
Other Study IDs: COMU-SBF-ME-01
Record Dates: First submitted 2024-05-02; First posted 2024-05-08 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Airway Complication of Anesthesia
Keywords: Airway Management; Ultrasonography; Pediatric Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laryngospasm and post-extubation stridor are major postoperative airway difficulties in pediatric patients using tracheal tubes. These conditions are frequently caused by epithelium edema and anesthesia-related problems. Because it could reveal tracheal and laryngeal issues, ultrasound is an essential method for establishing the proper endotracheal tube size and minimizing difficulties. This research focuses on the use of ultrasonography to predict and understand pediatric postoperative airway complications.

DETAILED DESCRIPTION:
In pediatric patients with tracheal tubes, laryngospasm, and post-extubation stridor are the two worst-case postoperative airway complications. Post-extubation stridor is caused by cricoid ring epithelial swelling, whereas laryngospasm is an uncommon but potentially fatal condition that occurs during the induction and recovery of anesthesia. When determining the proper endotracheal tube (ETT) size and minimizing postoperative problems, ultrasonography (USG) is important since it considers factors other than ETT size and irritation, like placement, surgical manipulation, and patient-specific circumstances. By displaying laryngeal and tracheal edema and the size and location of the ETT, ultrasound helps identify, at least in part, children who may experience respiratory issues. Thus, this research aims to illustrate how ultrasound could be utilized to predict the development of postoperative airway complications and to investigate the conditions that cause them in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1-11 years
* Anesthesia risk class: 1-2
* Patients who have given written consent

Exclusion Criteria:

* Patients aged under 1 or over 11 years
* Patients undergoing emergency surgery
* Patients with skin integrity issues such as open wounds, infections, or skin lesions in the area to be examined
* Patients with laryngeal or tracheal deformities
* Patients suspected of having a difficult airway
* Patients who have previously undergone surgery on the upper airway, larynx, or trachea
* Patients with a history of reactive airway disease (asthma, bronchial hyperreactivity)
* Patients who have had an upper respiratory tract infection within the last two weeks
* Patients with an anesthesia risk class of 3 or higher
* Patients undergoing high-risk surgery

Ages: 1 Year to 10 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients aged 1-11 years undergoing surgery under general anesthesia with an ASA classification of 1-2.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Association between Difference in Vocal Cord Thickness, and Postoperative Airway Complications | Vocal cord measurements are taken before intubation and extubation under general anesthesia, with complications assessed within the first hour postoperatively.
  This measure assesses the association between an increase in vocal cord thickness (measured in millimeters using ultrasonography) from pre-intubation to pre-extubation, and the incidence (%) of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction).
  Measurement Tool:
  * Ultrasonography to measure vocal cord thickness in millimeters.
  * The existence of post-operative airway complications is determined as follows: A post-operative airway complication is defined as cough, dysphonia, laryngospasm, or upper airway blockage within the first hour following surgery; if none of these findings are present, it is considered absent.
  Unit of Measure:
  * Millimeters for vocal cord thickness.
  * Categorical outcome (yes/no) for airway complications
Association between Difference in Subglottic Airway Wall Thickness, and Postoperative Airway Complications | Subglottic airway wall measurements are taken before intubation and extubation under general anesthesia, with complications assessed within the first hour postoperatively.
  This measure assesses the association between an increase in subglottic airway wall thickness (measured in millimeters using ultrasonography) from pre-intubation to pre-extubation, and the incidence (%) of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction).
  Measurement Tool:
  * Ultrasonography to measure subglottic airway wall thickness in millimeters.
  * The existence of post-operative airway complications is determined as follows: A post-operative airway complication is defined as cough, dysphonia, laryngospasm, or upper airway blockage within the first hour following surgery; if none of these findings are present, it is considered absent.
  Unit of Measure:
  * Millimeters for subglottic airway wall thickness.
  * Categorical outcome (yes/no) for airway complications

SECONDARY OUTCOMES:
Association Between Type of Surgery and Postoperative Airway Complications in Pediatric Patients | The type of surgery will be recorded at the preoperative examination, with airway complications assessed within the first hour postoperatively.
  This outcome measure assesses the association between different types of surgery (categorized by anatomical regions as head-neck, musculoskeletal, abdominal) and the occurrence of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction)
  Measurement Tool:
  * Classification of surgery type based on anatomical region. The classification will be as follows: 1st category head-neck, 2nd category abdomen, 3rd category musculoskeletal system surgeries.
  * The existence of post-operative airway complications is determined as follows: A post-operative airway complication is defined as cough, dysphonia, laryngospasm, or upper airway blockage within the first hour following surgery; if none of these findings are present, it is considered absent.
  Unit of Measure: Categorical (type of surgery); categorical outcome (presence/absence of airway complications).
Association Between the Difference in Outer Diameter of the Endotracheal Tube and the Narrowest Airway Diameter, and Postoperative Airway Complications | Airway and tube diameter measurements are taken intraoperatively before intubation under general anesthesia, with complications assessed within the first hour postoperatively.
  This measure assesses the association between the diffence between in the narrowest airway diameter the outer diameter of the endotracheal tube placed and the incidence (%) of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction)
  Measurement Tool:
  * Ultrasonography to measure the narrowest airway diameter.
  * The outer diameter of endotracheal tube measurement listed on the endotracheal tube packaging will be accepted.
  * The existence of post-operative airway complications is determined as follows: A post-operative airway complication is defined as cough, dysphonia, laryngospasm, or upper airway blockage within the first hour following surgery; if none of these findings are present, it is considered absent.
  Unit of Measure: Millimeters for airway and tube diameters; categorical outcome (presence/absence of airway complications).
Association Between Changes in Endotracheal Tube Position After Intubation and Before Extubation, and Postoperative Airway Complications | Measurements of endotracheal tube position are taken after intubation and before extubation under general anesthesia, with complications assessed within the first hour postoperatively
  This outcome measure evaluates the association between the change in the position of the endotracheal tube, as determined by ultrasonography after intubation and before extubation, and the incidence (%) of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction) Measurement Tool: Ultrasonography to assess changes in the position of the endotracheal tube.
  Unit of Measure:
  The endotracheal tube level will recorded as:
  Cricothyroid membrane, Cricoid cartilage, First tracheal cartilage, Second tracheal cartilage, Third and the other tracheal cartilages If the tube level has changed, it will be recorded as 'change present'; if it remains the same, it will be recorded as 'no change'.
  Position changes are categorical (change/no change); complications are categorical outcomes(presence/absence of airway complications).
Association Between Endotracheal Tube Position Before Extubation and Postoperative Airway Complications | Endotracheal tube position is recorded before extubation intraoperatively under general anesthesia, with complications assessed within the first hour postoperatively
  : This outcome measure assesses the association between the endotracheal tube position before extubation, as determined by ultrasonography, and the incidence (%) of postoperative airway complications (categorical: presence or absence of cough, dysphonia, symptom of laryngospasm, and sign of upper airway obstruction)
  Measurement Tool: Ultrasonography to measure the position of the endotracheal tube.
  Unit of Measure: Tube position is categorized based on anatomical landmarks (1st category, 2nd category cricothyroid membrane, 3 rd category cricoid cartilage, 4 th category first tracheal cartilage, 5 th category second tracheal cartilage, 6 th category third and other tracheal cartilages); complications are categorical outcomes (presence/absence of airway complications).

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Çanakkale, Turkey (Türkiye)